CLINICAL TRIAL: NCT03342131
Title: Change of Serum Wnt2 or Wnt4 and the Relationship With Hs-CRP，cTnI and Prognosis in Patients With Acute Coronary Syndrome
Brief Title: Serum Concentration of Wnt2 and Wnt4 in Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: PJ-KS-KY-2017-104(X)
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2017-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Wnt signaling
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- STEMI group: The study population consists of 150 patients with ST-elevated acute myocardial infarction (STEMI) who are admitted within 24 hours after chest pain attack. They will all undergo coronary angiography. The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, asthma, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded. Blood (150 each group) is obtained into ethylenediaminetetraacetic acid（EDTA） tubes from all subjects via antecubital venepuncture to explore circulating wnt 2 and wnt 4 concentration by ELISA at 0 , 7days and 12 months after admission.
  Interventions: Other: Circulating wnt 2 and wnt 4 concentration
- NST-ACS group: The study population consists of 150 patients with non-ST elevated acute myocardial infarction (NST-ACS) including unstable angina pectoris (UAP),who are admitted within 24 hours after chest pain attack. They will all undergo coronary angiography. The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, asthma, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded.Blood (150 each group) is obtained into ethylenediaminetetraacetic acid（EDTA） tubes from all subjects via antecubital venepuncture to explore circulating wnt 2 and wnt 4 concentration by ELISA at 0 , 7days and 12 months after admission.
  Interventions: Other: Circulating wnt 2 and wnt 4 concentration
- Control group: 150 age and body mass index matched healthy subjects with neither coronary artery disease nor any of the components of the metabolic syndrome are studied as Control group. Circulation wnt2 and wnt4 concentration in Control group will be measured only once with 24h after admission.
  Interventions: Other: Circulating wnt 2 and wnt 4 concentration

INTERVENTIONS:
Other: Circulating wnt 2 and wnt 4 concentration — Blood (150 each group) is obtained into ethylenediaminetetraacetic acid（EDTA） tubes from all subjects via antecubital venepuncture to explore circulating wnt 2 and wnt 4 concentration by ELISA. Continuous wnt2 and wnt4 concentration are measured in all patients with STEMI at 0 , 7days and 12 months after admission. Other patients with acute syndrome system are measured Wnt 2 and wnt4 only once within 24h after admission.
  Wnt2 and wnt4 concentration in Control group will be measured only once with 24h after admission.

SUMMARY:
This study aims to find the change of serum wnt effectory moleculars and the association with Hs-CRP，cTnI and Prognosis in Patients with Acute Coronary Syndrome.

DETAILED DESCRIPTION:
It has been reported that wnt effecory moleculars (wnt2, wnt4, wnt11,wnt10b, DKK1, DKK2) increased in myocardium at acute phase after myocardium infarction in animal experiment. These moleculars can be detected in serum or plasma from human subjects. However, there is few relevant studies about wnt2 and wnt4 concentration in patients with acute coronary syndrome. This study valuates the serum wnt2 and wnt4 concentration in patients with acute coronary syndrome. It will possibly enable to find the relationship between serum wnt2 or wnt4 concentration and Hs-CRP, cTnI and prognosis in patients with Acute Coronary Syndrome.

ELIGIBILITY:
Inclusion Criteria:

.diagnosed as acute coronary syndrome, including STEMI and NST-ACS.

* with left ventricular ejection fraction（LVEF）>=45%
* written informed consents are obtained
* admitted within 24 hours after chest pain attacked

Exclusion Criteria:

* • complicated with rheumatic heart disease, coronary arteritis, hypertrophic cardiomyopathy or dilated cardiomyopathy

  * complicated with malignant tumor,the immune system diseases, blood system diseases, recently (within 2 weeks) taking glucocorticoid drugs, the use of immunosuppressive agents and cerebral infarction
  * with acute or chronic infection, surgery or trauma in the last month
  * secondary hypertension, severe liver dysfunction,severe renal insufficiency
  * with abnormal thyroid function or allergy to iodine agent refusal to sign the informed consent

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome,including STEMI and NST-ACS group patients
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-09-29 (Estimated); Study Completion 2019-03-29 (Estimated)

PRIMARY OUTCOMES:
Serum wnt2 and wnt4 concentration | 12 months
  Serum wnt2 and wnt4 concentration in ng/ml

SECONDARY OUTCOMES:
Relationship between wnt2 or wnt4 and high sensitive C reaction protein (hs-CRP) concentration | 12 months
  Correlation of wnt2 and wnt4 with hs-CRP concentration
Relationship between wnt2 or wnt4 and Troponin-I (Tn-I) concentration | 12 months
  Correlation of wnt2 and wnt4 with Tn-I concentration
MACEs during 12-month follow-up | 12 months
  Association of wnt2 or wnt4 concentration with prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Rongchong Huang, Ph,D, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
We will publish the paper to described the data and share with other researchers

REFERENCES:
- [Result] Aisagbonhi O, Rai M, Ryzhov S, Atria N, Feoktistov I, Hatzopoulos AK. Experimental myocardial infarction triggers canonical Wnt signaling and endothelial-to-mesenchymal transition. Dis Model Mech. 2011 Jul;4(4):469-83. doi: 10.1242/dmm.006510. Epub 2011 Feb 14. PMID 21324930
- [Result] Perez Castrillon JL, San Miguel A, Vega G, Abad L, Andres Domingo M, Gonzalez Sagredo M, de Luis D, Duenas-Laita A. Levels of DKK1 in patients with acute myocardial infarction and response to atorvastatin. Int J Cardiol. 2010 Nov 5;145(1):164-5. doi: 10.1016/j.ijcard.2009.07.025. Epub 2009 Aug 31. PMID 19720407
- [Result] Wang L, Hu XB, Zhang W, Wu LD, Liu YS, Hu B, Bi CL, Chen YF, Liu XX, Ge C, Zhang Y, Zhang M. Dickkopf-1 as a novel predictor is associated with risk stratification by GRACE risk scores for predictive value in patients with acute coronary syndrome: a retrospective research. PLoS One. 2013;8(1):e54731. doi: 10.1371/journal.pone.0054731. Epub 2013 Jan 24. PMID 23359112
- [Result] Alexandrovich A, Arno M, Patient RK, Shah AM, Pizzey JA, Brewer AC. Wnt2 is a direct downstream target of GATA6 during early cardiogenesis. Mech Dev. 2006 Apr;123(4):297-311. doi: 10.1016/j.mod.2006.02.002. Epub 2006 Apr 18. PMID 16621466
- [Result] Caprioli A, Villasenor A, Wylie LA, Braitsch C, Marty-Santos L, Barry D, Karner CM, Fu S, Meadows SM, Carroll TJ, Cleaver O. Wnt4 is essential to normal mammalian lung development. Dev Biol. 2015 Oct 15;406(2):222-34. doi: 10.1016/j.ydbio.2015.08.017. Epub 2015 Aug 29. PMID 26321050
- [Result] Goodwin AM, D'Amore PA. Wnt signaling in the vasculature. Angiogenesis. 2002;5(1-2):1-9. doi: 10.1023/a:1021563510866. PMID 12549854